CLINICAL TRIAL: NCT05733221
Title: Determining the Ease of Utilizing 3D Printed Models to Aide in Isolated Mandibular Fracture Repair
Brief Title: 3D Printed Models for Mandibular Fracture Repair
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Deepak Krishnan, Chief of Oral & Maxillofacial Surgery, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0794
Record Dates: First submitted 2023-01-10; First posted 2023-02-17 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Mandible Fracture; Maxillofacial Trauma
Keywords: 3D Printing; Personalized Medicine; Maxillofacial Trauma
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Intervention Model Description: The investigators propose a parallel design randomized control trial to study the value of 3D printing for preoperative planning in patients with a fracture of the mandible who require open reduction, internal fixation. The study will be split into two arms: 1) Patients that will have a 3D model generated for the surgical procedure 2) The control group who will follow normal standards of care as outlined above and won't have the additional 3D model created pre-operatively.
Who Masked: Participant
Masking Description: Once the subjects are identified the research coordinator will conduct a screening of the patient to ensure they meet the inclusion/ exclusion criteria for the study and then randomize the patient into either normal standard of care for surgical repair of the fractured mandible or normal standard of care for surgical repair of the fractured mandible aided by a 3D printed model of the patient's jaw.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- 3D Model Generated (Experimental): Patient will undergo an Open Reduction and Internal Fixation preformed by a surgeon who had pre-operative access to a 3D model printed to help pre-bend hardware.
  Interventions: Device: 3D Printed Model
- Normal Standards of Care without Aide of Model (No Intervention): Patient will undergo standard Open Reduction and Internal Fixation by a surgeon who did not have a pre-operative 3D model.

INTERVENTIONS:
Device: 3D Printed Model — 3D Printed Model generated pre-operatively of the patients mandible.
  Arms: 3D Model Generated

SUMMARY:
The investigators will test the hypothesis that patients randomized to the intervention (3D printing with pre-bent plate) arm have less operative room time and less time for the critical part of the procedure than patients in the control arm (no 3D printing, current standards of care). Personalized medicine and care for fracture treatment.

DETAILED DESCRIPTION:
The goal of treatment is to re-establish the patient's preinjury dental occlusion and facial harmony. Fractures that are nondisplaced and exhibit no occlusal changes may be amenable to nonsurgical management, but most mandible fractures will require stabilization for satisfactory healing and to restore pretraumatic maxillomandibular orientation. Various treatment strategies have been described and vary widely depending on the fracture location and surgeon's preference. The patient's demographics, comorbidities, dentition, and fracture characterization will all influence the choice of fixation by the treating surgeon.

There are very few randomized control trials that show outcomes when 3D printing is used for intervention planning and performing a procedure. These data are essential to establish value of 3D printing as a clinical service. There is also anecdotal evidence that a 3D printed model of a mandible fracture can be useful for pre-operative planning because the oral and maxillofacial surgeon can better assess the geometry of the bone lesions and can pre-bend fixation plates before the procedure. This hypothetically decreases the amount of time in the operating room.

The investigators propose a parallel design randomized control trial to study the value of 3D printing for preoperative planning in patients with a fracture of the mandible who require open reduction, internal fixation. The study will be split into two arms: 1) Patients that will have a 3D model generated for the surgical procedure 2) The control group who will follow normal standards of care as outlined above and won't have the additional 3D model created pre-operatively.

ELIGIBILITY:
Inclusion Criteria:

Patient ≥ 18 years of age

* Patients who have received either a cone beam or conventional CT
* Admitted through University of Cincinnati Hospital and Medical Center emergency department
* All isolated mandible fractures referred to University of Cincinnati Hospital Oral & maxillofacial surgery clinic
* Surgical team members from the division of plastic and otolaryngology

Exclusion Criteria:

* Patient < 18 years of age
* Patients who have neither cone beam nor conventional CT
* Patients requiring a repeat procedure
* Unexpected exposure of hardware

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total time in the OR | Total procedural time
  Time in the OR considered critical part of the procedure by the Oral & Maxillofacial Surgery Staff
Subjective outcome to surgeon | Up to 2 days post-procedure
  Surgeon overall satisfaction with utilizing the 3D generated model, obtained via Likert Scale Questions completed post-operatively. The investigators are going to use the Likert questions to develop a numerical scoring system and report that data as "raw" Likert scores. Likert questions and conversion of specialists' responses to Anatomic Model Utility Points (AMUPs). Responses of "strongly disagree", "disagree", and "neutral" were assigned 0 AMUP points. Responses to preprocedural confidence are assigned negative points, to effectively subtract the impact of the anatomic model post- versus pre-procedure. The maximum AMUP for each patient was 500.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak G Krishnan, DDS, Principal Investigator — University of Cincinnati
Locations (2):
- United States (2):
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UC Health Holmes Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Background] de Vries EN, Ramrattan MA, Smorenburg SM, Gouma DJ, Boermeester MA. The incidence and nature of in-hospital adverse events: a systematic review. Qual Saf Health Care. 2008 Jun;17(3):216-23. doi: 10.1136/qshc.2007.023622. PMID 18519629
- [Background] Visser A, Geboers B, Gouma DJ, Goslings JC, Ubbink DT. Predictors of surgical complications: A systematic review. Surgery. 2015 Jul;158(1):58-65. doi: 10.1016/j.surg.2015.01.012. Epub 2015 Feb 27. PMID 25731783
- [Background] Cheng H, Clymer JW, Po-Han Chen B, Sadeghirad B, Ferko NC, Cameron CG, Hinoul P. Prolonged operative duration is associated with complications: a systematic review and meta-analysis. J Surg Res. 2018 Sep;229:134-144. doi: 10.1016/j.jss.2018.03.022. Epub 2018 Apr 24. PMID 29936980
- [Background] Adi M, Ogden GR, Chisholm DM. An analysis of mandibular fractures in Dundee, Scotland (1977 to 1985). Br J Oral Maxillofac Surg. 1990 Jun;28(3):194-9. doi: 10.1016/0266-4356(90)90088-3. PMID 2135661
- [Background] Telfer MR, Jones GM, Shepherd JP. Trends in the aetiology of maxillofacial fractures in the United Kingdom (1977-1987). Br J Oral Maxillofac Surg. 1991 Aug;29(4):250-5. doi: 10.1016/0266-4356(91)90192-8. PMID 1911673
- [Background] Chrcanovic BR, Abreu MH, Freire-Maia B, Souza LN. 1,454 mandibular fractures: a 3-year study in a hospital in Belo Horizonte, Brazil. J Craniomaxillofac Surg. 2012 Feb;40(2):116-23. doi: 10.1016/j.jcms.2011.03.012. Epub 2011 Mar 31. PMID 21458284
- [Background] Pickrell BB, Serebrakian AT, Maricevich RS. Mandible Fractures. Semin Plast Surg. 2017 May;31(2):100-107. doi: 10.1055/s-0037-1601374. PMID 28496390
- [Background] AO Foundation. AO Surgery reference. Available at: https://www2.aofoundation.org/.
- [Background] Ellis E 3rd, Miles BA. Fractures of the mandible: a technical perspective. Plast Reconstr Surg. 2007 Dec;120(7 Suppl 2):76S-89S. doi: 10.1097/01.prs.0000260721.74357.e7. PMID 18090731
- [Background] Nishioka GJ, Van Sickels JE. Transoral plating of mandibular angle fractures: a technique. Oral Surg Oral Med Oral Pathol. 1988 Nov;66(5):531-5. doi: 10.1016/0030-4220(88)90370-2. PMID 3200555
- [Background] Ellis E 3rd. A study of 2 bone plating methods for fractures of the mandibular symphysis/body. J Oral Maxillofac Surg. 2011 Jul;69(7):1978-87. doi: 10.1016/j.joms.2011.01.032. Epub 2011 May 6. PMID 21549485
- [Background] Agnihotri A, Prabhu S, Thomas S. A comparative analysis of the efficacy of cortical screws as lag screws and miniplates for internal fixation of mandibular symphyseal region fractures: a randomized prospective study. Int J Oral Maxillofac Surg. 2014 Jan;43(1):22-8. doi: 10.1016/j.ijom.2013.07.001. Epub 2013 Aug 6. PMID 23928155
- [Background] King BJ, Park EP, Christensen BJ, Danrad R. On-Site 3-Dimensional Printing and Preoperative Adaptation Decrease Operative Time for Mandibular Fracture Repair. J Oral Maxillofac Surg. 2018 Sep;76(9):1950.e1-1950.e8. doi: 10.1016/j.joms.2018.05.009. Epub 2018 May 15. PMID 29859953
- [Background] Furr AM, Schweinfurth JM, May WL. Factors associated with long-term complications after repair of mandibular fractures. Laryngoscope. 2006 Mar;116(3):427-30. doi: 10.1097/01.MLG.0000194844.87268.ED. PMID 16540903
- [Background] Senel FC, Jessen GS, Melo MD, Obeid G. Infection following treatment of mandible fractures: the role of immunosuppression and polysubstance abuse. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Jan;103(1):38-42. doi: 10.1016/j.tripleo.2006.02.013. Epub 2006 Aug 10. PMID 17178492
- [Background] Odono, Lauren, et al. "Mandible Fractures." Facial Trauma Surgery, 14th ed., vol. 1, Elsevier, Amsterdam, Netherlands, 2020, pp. 168-185.
- [Background] Bochlogyros PN. Non-union of fractures of the mandible. J Maxillofac Surg. 1985 Aug;13(4):189-93. doi: 10.1016/s0301-0503(85)80046-1. PMID 3860599
- [Background] Melmed EP, Koonin AJ. Fractures of the mandible. A review of 909 cases. Plast Reconstr Surg. 1975 Sep;56(3):323-7. doi: 10.1097/00006534-197509000-00011. PMID 239432
- [Background] Ogasawara T, Sano K, Hatsusegawa C, Miyauchi K, Nakamura M, Matsuura H. Pathological fracture of the mandible resulting from osteomyelitis successfully treated with only intermaxillary elastic guiding. Int J Oral Maxillofac Surg. 2008 Jun;37(6):581-3. doi: 10.1016/j.ijom.2007.11.006. Epub 2008 Feb 12. PMID 18272342
- [Background] Quadu G, Miotti A, Rubini L. [Chronic osteomyelitis of the mandible with pathologic fracture. Case report]. G Stomatol Ortognatodonzia. 1983 Jul-Sep;2(3):99-100. No abstract available. Italian. PMID 6590496
- [Background] Jauhar P, Handley T, Hammersley N. A Pathological Fracture of the Mandible due to Osteomyelitis following a Full Dental Clearance. Dent Update. 2016 Mar;43(2):168-70, 173, 175. doi: 10.12968/denu.2016.43.2.168. PMID 27188132
- [Background] Wagner WF, Neal DC, Alpert B. Morbidity associated with extraoral open reduction of mandibular fractures. J Oral Surg. 1979 Feb;37(2):97-100. PMID 283211
- [Background] Mehra P, Murad H. Internal fixation of mandibular angle fractures: a comparison of 2 techniques. J Oral Maxillofac Surg. 2008 Nov;66(11):2254-60. doi: 10.1016/j.joms.2008.06.024. PMID 18940489
- [Background] Ravi P, Burch MB, Farahani S, Chepelev LL, Yang D, Ali A, Joyce JR, Lawera N, Stringer J, Morris JM, Ballard DH, Wang KC, Mahoney MC, Kondor S, Rybicki FJ; University of Cincinnati 3D Printing Clinical Service Participants. Utility and Costs During the Initial Year of 3D Printing in an Academic Hospital. J Am Coll Radiol. 2023 Feb;20(2):193-204. doi: 10.1016/j.jacr.2022.07.001. Epub 2022 Aug 18. PMID 35988585

DOCUMENTS (2):
  • Study Protocol (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT05733221/Prot_000.pdf
  • Informed Consent Form (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT05733221/ICF_001.pdf